CLINICAL TRIAL: NCT05338736
Title: Differences in Humoral and Cellular Immunity in First-cycle Vaccinated Patients Infected by SARS-COV-2: an Observational Study
Brief Title: Humoral and Cellular Immunity in First-cycle SARS-CoV-2 Vaccinated COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Director of the Intensive Care and Anesthesia Department, University Magna Graecia
Other Study IDs: Immune-COVID
Record Dates: First submitted 2022-04-19; First posted 2022-04-21 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: SARS CoV 2 Infection; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Twenty milliliters of whole blood will be collected from every included patient. Two milliliters will be centrifuged to obtain plasma within a speed range of 1300-2000g, for 10min at 25 ° C. Eighteen milliliters will be subjected to Ficoll density gradient separation to isolate mononuclear cells (PBMCs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Control patients with a complete first-cycle vaccination against SARS-CoV-2, received between 4 to 7 months before the inclusion, and with a nasopharyngeal swab negative for SARS-CoV-2 isolation.
  Interventions: Diagnostic Test: LIAISON SARS-CoV-2 TrimericS IgG (DiaSorin); Diagnostic Test: LIAISON SARS-CoV2-IgM (DiaSorin); Diagnostic Test: Human IFN-g ELISpot PLUS (ALP) (AUROGENE)
- Asymptomatic group: Patients with a complete first-cycle vaccination against SARS-CoV-2, received between 4 to 7 months before the inclusion, with a nasopharyngeal swab positive for SARS-CoV-2 isolation, in absence of any symptoms of COVID-19
  Interventions: Diagnostic Test: LIAISON SARS-CoV-2 TrimericS IgG (DiaSorin); Diagnostic Test: LIAISON SARS-CoV2-IgM (DiaSorin); Diagnostic Test: Human IFN-g ELISpot PLUS (ALP) (AUROGENE)
- Symptomatic group: Patients with a complete first-cycle vaccination against SARS-CoV-2, received between 4 to 7 months before the inclusion, with a nasopharyngeal swab positive for SARS-CoV-2 isolation, with moderate to severe symptoms of COVID-19
  Interventions: Diagnostic Test: LIAISON SARS-CoV-2 TrimericS IgG (DiaSorin); Diagnostic Test: LIAISON SARS-CoV2-IgM (DiaSorin); Diagnostic Test: Human IFN-g ELISpot PLUS (ALP) (AUROGENE)

INTERVENTIONS:
Diagnostic Test: LIAISON SARS-CoV-2 TrimericS IgG (DiaSorin) — Kit to test the concentration of Immunoglobulin G anti-SARS-CoV-2 in the plasma of included patients
Diagnostic Test: LIAISON SARS-CoV2-IgM (DiaSorin) — Kit to test the concentration of Immunoglobulin M anti-SARS-CoV-2 in the plasma of included patients
Diagnostic Test: Human IFN-g ELISpot PLUS (ALP) (AUROGENE) — Kit to test the cellular immunity response by measuring the Interferon gamma released by mononuclear cells (PBMCs)

SUMMARY:
Infection by the recent Coronavirus (SARS-CoV-2) has generated at a pandemic level a new pathology, called COVID-19, characterized by "flu-like" symptoms up to severe acute respiratory failure. The pathogenesis of the disease involves both humoral and cellular immunological responses; cell-mediated immunity is the first and most effective immune response to viral infection. To date, despite the extensive scientific research aimed at curing COVID-19, there are few effective means to tackle SARS-CoV-2 infection and reduce its disease progression. Among these, a first complete anti-SARS-CoV-2 vaccination course has been shown to significantly reduce the development of the disease towards the more severe forms requiring hospital and intensive care. On the other hand, over time the antibody response induced by vaccines against SARS-CoV-2 decreases, so much so as to indicate the need for a third booster dose. This translates into the fact that some patients who have undergone a complete first vaccination course, with third dose booster indications, develop severe critical disease, with the need for hospitalization. On the other hand, other patients with the same vaccination status do not develop the disease, although they are also positive for SARS-CoV-2. The investigators therefore hypothesized that the humoral and cell-mediated response among groups of patients may be radically different. For these reasons, the investigators designed this observational pilot study in order to analyze humoral and cell-mediated responses in SARS-CoV-2 positive first complete vaccination patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a complete first-cycle vaccination against SARS-CoV-2 performed 4 to 7 months before.

Exclusion Criteria:

* Presence of malignancy under chemotherapy
* Patient with previous transplantation
* Patient receiving immuno-modulatory or immunosuppressive drugs
* Patient receiving corticosteroid therapy since more than 10 days
* Pregnancy
* Consent withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Forty-five patients will be totally enrolled in the study. Three cohorts of patients will be considered.
  1. Control group: 15 vaccinated patients with a pharyngeal swab negative for SARS-CoV-2 isolation
  2. Asymptomatic group: 15 vaccinated patients with a pharyngeal swab positive for SARS-CoV-2 isolation and absence of symptoms related to the infection
  3. Symptomatic group: 15 vaccinated patients with a pharyngeal swab positive for SARS-CoV-2 isolation and presence of moderate to severe symptoms related to the infection (i.e. peripheral oxygen saturation lower than 94% in room air)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Differences between populations with respect to anti-SARS-CoV-2 immunoglobulins | At day 0
  After obtaining plasma of included patients, the plasma will be processed with a dedicated kit to measure the concentration of Immunoglobulin G and M. Differences between patients' cohorts will be assessed
Differences between populations with respect to cellular immunity | At day 0
  Mononuclear immunity cells will be analyzed with a dedicated ELISpot kit to assess their response to SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Principal Investigator — Magna Graecia University
Locations (1):
- AOU Mater Domini, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
The individual patients data will be shared only after the publication of the study on an international peer-reviewed journal and on scientific and intelligible proposal
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after publication on an indexed international and peer-reviewed journal
Access Criteria: Access will be allowed after contacting by email the principal investigator, by providing and intelligible and scientific proposal